CLINICAL TRIAL: NCT03923738
Title: A Phase Ib, Open-Label, Dose-Ranging Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Tocilizumab Administered by Intravenous Infusion to Patients With Giant Cell Arteritis
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Tocilizumab (TCZ) Administered to Participants With Giant Cell Arteritis (GCA).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP41152; 2018-004718-17 (EudraCT Number)
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TCZ IV Q4W (Experimental): Participants will receive up to 6 doses of Dose 1 of TCZ IV Q4W followed by up to 6 doses of Dose 2 of TCZ IV Q4W.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — TCZ will be administered by IV infusion at two dose levels Q4W. The maximum dose of TCZ that will be administered is 800 mg. The dose of TCZ infusion will be calculated on the basis of body weight measured prior to each infusion.
  Other Names: RoActemra/Actemra

SUMMARY:
This study will evaluate the pharmacokinetics, pharmacodynamics, and safety of two dose levels of tocilizumab (TCZ) administered by intravenous (IV) infusion every 4 weeks (Q4W) to participants with giant cell arteritis (GCA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA as classified according to protocol-specified criteria;
* Participants entering Period 1 must be receiving treatment with TCZ 8 mg/kg IV Q4W.

Exclusion Criteria:

* Treatment with any other investigational agent besides TCZ within 12 weeks (or 5 half-lives of the investigational drug, whichever is longer) prior to screening;
* Evidence of serious uncontrolled disease;
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections;
* Active TB requiring treatment within the previous 3 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Switzerland (2):
  - Universitätsspital Basel; Rheumatologie, Basel
  - Inselspital Bern; Rheumatologie; Klinische Immunologie und Allergologie, Bern

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Schmitt C, Brockwell L, Giraudon M, Zucchetto M, Christ L, Bannert B, Daikeler T, Villiger PM. Intravenous tocilizumab for the treatment of giant cell arteritis: a phase Ib dose-ranging pharmacokinetic bridging study. Arthritis Res Ther. 2022 Jun 4;24(1):133. doi: 10.1186/s13075-022-02815-9. PMID 35659282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from Period 1 (n=24) that completed the Period and reached remission entered Period 2 (n=22). Two participants withdrew prior to entering Period 2.
Groups:
- TCZ IV Q4W: Participants with GCA who received at least 5 consecutive doses of 8 mg/kg IV TCZ Q4W prior to baseline and reached remission received 5 or 6 consecutive doses of 7 mg/kg IV TCZ Q4W in Period 1. Participants that completed Period 1 and were in remission received 5 or 6 consecutive doses of 6 mg/kg IV TCZ Q4W in Period 2.
Period: Period 1
Arm/Group | TCZ IV Q4W
Started | 24
Completed | 22
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2
Arm/Group | TCZ IV Q4W
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TCZ IV Q4W
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of TCZ
Time Frame: Baseline; Weeks 4, 8, 12, 16-24
Population: The pharmacokinetic (PK) population consisted of participants who received one dose of TCZ and had one valid PK sample, with participants grouped according to treatment received.
Measure: Median (Full Range); unit: ug/mL
Groups:
- TCZ IV Q4W 7 mg/kg: Participants with GCA who received at least 5 consecutive doses of 8 mg/kg TCZ prior to baseline and reached remission received 5 or 6 consecutive doses of 7 mg/kg IV TCZ Q4W (Period 1).
- TCZ IV Q4W 6 mg/kg: Participants that completed Period 1 and were in remission received 5 or 6 consecutive doses of 6 mg/kg IV TCZ Q4W (Period 2).
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 21 | 22
ug/mL | 197 [118 to 352] | 178 [115 to 320]

2. Primary Outcome: Trough Serum Concentration (Ctrough) of TCZ at Steady State
Time Frame: Baseline; Weeks 4, 8, 12, 16-24
Population: as for outcome 1
Measure: Median (Full Range); unit: ug/mL
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 22 | 22
ug/mL | 37.2 [6.59 to 69.0] | 22.7 [3.38 to 54.5]

3. Primary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval of 4 Weeks (AUC4weeks) of TCZ at Steady State
Time Frame: Baseline; Weeks 4, 8, 12, 16-24
Population: as for outcome 1
Measure: Median (Full Range); unit: day*ug/mL
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 22 | 22
day*ug/mL | 2130 [1120 to 4300] | 1610 [921 to 3070]

4. Primary Outcome: Percentage of Participants With Adverse Events
Time Frame: Baseline - Day 151
Measure: Number; unit: Percentage of Participants
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 24 | 22
Percentage of Participants | 79.2 | 40.9

5. Secondary Outcome: Serum Concentration of Interleukin-6 (IL-6)
Time Frame: Baseline; Weeks 12, 16, 20, 24
Population: The pharmacodynamic (PD) population was identical to the safety analysis population, which consisted of participants who received at least one dose of study drug and had at least one safety assessment.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 24 | 22
pg/mL
  Baseline: number analyzed (Participants) | 24 | 20
  Baseline | 57.80 (61.149) | 39.46 (25.989)
  Week 12: number analyzed (Participants) | 22 | 21
  Week 12 | 56.03 (84.988) | 49.73 (81.718)
  Week 16: number analyzed (Participants) | 22 | 21
  Week 16 | 97.57 (277.409) | 43.04 (54.232)
  Week 20: number analyzed (Participants) | 22 | 21
  Week 20 | 38.11 (21.147) | 46.97 (61.454)
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 111.00 (NA) — SD is NA for n=1 |

6. Secondary Outcome: Serum Concentration of Soluble Interleukin-6 Receptor (sIL-6R)
Time Frame: Baseline; Weeks 12, 16, 20, 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 24 | 22
ng/mL
  Baseline: number analyzed (Participants) | 24 | 20
  Baseline | 665.8 (153.81) | 671.3 (152.69)
  Week 12: number analyzed (Participants) | 22 | 21
  Week 12 | 680.8 (183.84) | 670.9 (175.92)
  Week 16: number analyzed (Participants) | 22 | 21
  Week 16 | 654.6 (173.26) | 651.7 (136.95)
  Week 20: number analyzed (Participants) | 22 | 21
  Week 20 | 663.8 (147.92) | 690.0 (215.91)
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 519.0 (NA) — SD is NA for n=1 |

7. Secondary Outcome: Serum Concentration of C-Reactive Protein (CRP)
Time Frame: Baseline; Weeks 4, 8, 12, 16-24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 24 | 22
mg/L
  Baseline | 0.615 (1.1645) | 0.356 (0.2486)
  Week 4: number analyzed (Participants) | 22 | 22
  Week 4 | 0.511 (0.7538) | 0.591 (1.0646)
  Week 8: number analyzed (Participants) | 23 | 22
  Week 8 | 0.426 (0.3687) | 0.403 (0.3217)
  Week 12: number analyzed (Participants) | 23 | 22
  Week 12 | 0.467 (0.5694) | 0.359 (0.2585)
  Week 16: number analyzed (Participants) | 21 | 20
  Week 16 | 0.344 (0.2795) | 0.382 (0.3726)
  Week 17: number analyzed (Participants) | 19 | 22
  Week 17 | 0.409 (0.2533) | 0.409 (0.4521)
  Week 18: number analyzed (Participants) | 19 | 22
  Week 18 | 0.374 (0.2994) | 0.389 (0.3168)
  Week 19: number analyzed (Participants) | 19 | 21
  Week 19 | 0.387 (0.2801) | 0.388 (0.3348)
  Week 20: number analyzed (Participants) | 19 | 20
  Week 20 | 0.340 (0.2172) | 0.416 (0.2938)
  Week 21: number analyzed (Participants) | 2 | 0
  Week 21 | 0.200 (0.0000) |
  Week 22: number analyzed (Participants) | 3 | 0
  Week 22 | 0.200 (0.0000) |
  Week 23: number analyzed (Participants) | 3 | 0
  Week 23 | 0.203 (0.0058) |
  Week 24: number analyzed (Participants) | 3 | 0
  Week 24 | 0.200 (0.0000) |

8. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Time Frame: Baseline; Weeks 4, 8, 12, 16-24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | TCZ IV Q4W 7 mg/kg | TCZ IV Q4W 6 mg/kg
Number analyzed (Participants) | 24 | 22
mm/h
  Baseline | 6.1 (6.72) | 5.6 (5.01)
  Week 4: number analyzed (Participants) | 22 | 22
  Week 4 | 4.7 (3.38) | 5.6 (4.11)
  Week 8: number analyzed (Participants) | 23 | 22
  Week 8 | 7.2 (12.25) | 5.0 (3.13)
  Week 12: number analyzed (Participants) | 23 | 22
  Week 12 | 5.9 (5.30) | 6.5 (5.27)
  Week 16: number analyzed (Participants) | 21 | 20
  Week 16 | 5.9 (4.56) | 5.1 (4.32)
  Week 17: number analyzed (Participants) | 19 | 22
  Week 17 | 5.2 (3.84) | 5.0 (4.64)
  Week 18: number analyzed (Participants) | 19 | 22
  Week 18 | 4.4 (3.99) | 4.8 (3.01)
  Week 19: number analyzed (Participants) | 19 | 21
  Week 19 | 4.3 (2.64) | 5.0 (5.20)
  Week 20: number analyzed (Participants) | 19 | 20
  Week 20 | 7.1 (6.19) | 5.6 (5.04)
  Week 21: number analyzed (Participants) | 2 | 0
  Week 21 | 4.5 (3.54) |
  Week 22: number analyzed (Participants) | 3 | 0
  Week 22 | 5.3 (3.79) |
  Week 23: number analyzed (Participants) | 3 | 0
  Week 23 | 4.0 (3.00) |
  Week 24: number analyzed (Participants) | 3 | 0
  Week 24 | 3.7 (1.53) |

ADVERSE EVENTS:
Time Frame: Baseline - Day 151
Groups:
- TCZ IV 7 mg/kg Q4W: Participants with GCA who received at least 5 consecutive doses of 8 mg/kg TCZ prior to baseline and reached remission received 5 or 6 consecutive doses of 7 mg/kg IV TCZ Q4W (Period 1).
- TCZ IV 6 mg/kg Q4W: Participants that completed Period 1 and were in remission received 5 or 6 consecutive doses of 6 mg/kg IV TCZ Q4W (Period 2).
Arm/Group | TCZ IV 7 mg/kg Q4W | TCZ IV 6 mg/kg Q4W
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/22
Other Adverse Events (participants affected / at risk) | 6/24 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCZ IV 7 mg/kg Q4W (N=24) | TCZ IV 6 mg/kg Q4W (N=22)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCZ IV 7 mg/kg Q4W (N=24) | TCZ IV 6 mg/kg Q4W (N=22)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03923738/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03923738/SAP_001.pdf